CLINICAL TRIAL: NCT02994082
Title: Treating Smokeless Tobacco Use in Rural Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mark Vander Weg (U.S. Federal Agency)
Collaborators: Iowa City VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Mark Vander Weg, Reserach Specialist, Iowa City Veterans Affairs Medical Center
Organization: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201611737
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Smokeless Tobacco; Nicotine Dependence
Keywords: Rural health; Veterans; Smokeless tobacco cessation
MeSH Terms: conditions — Tobacco Use; Tobacco Use Disorder; Tobacco Use Cessation | interventions — Ethanol; Tobacco Use Cessation Devices; Nicotine Chewing Gum; Bupropion; Varenicline; Health Records, Personal; Contraindications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Intervention (Experimental): The tailored behavioral intervention includes both behavioral and pharmacological components. The behavioral component will consist of six sessions of cognitive behavioral therapy and coping skills training delivered over the telephone. In addition, participants will be screened for conditions commonly associated with tobacco use (depressive symptoms, risky alcohol use, weight concerns) and offered supplementary behavioral treatment modules to address these issues. Participants will also be offered pharmacotherapy for tobacco cessation, with decisions regarding specific medication(s) based on patients' medical history, contraindications, prior experiences, and preferences.
  Interventions: Behavioral: Tailored behavioral intervention; Behavioral: Behavioral activation for elevated depressive symptoms; Behavioral: Post-cessation weight gain management; Behavioral: Alcohol use risk reduction; Drug: Nicotine replacement therapy - transdermal nicotine patch; Drug: Nicotine replacement therapy - nicotine lozenge; Drug: Nicotine replacement therapy - nicotine gum; Drug: Bupropion sustained release; Drug: Varenicline; Drug: Combination nicotine replacement therapy; Drug: Combination nicotine replacement therapy + bupropion
- Facilitated tobacco quit line referral (Active Comparator): Participants assigned to this condition will receive information about the VA telephone tobacco quit line and educational materials and encouraged to enroll in treatment. In addition, they will be given information regarding available medications for smoking cessation and encouraged to contact their primary care provider to discuss their options.
  Interventions: Behavioral: Tobacco quit line; Behavioral: Educational materials

INTERVENTIONS:
Behavioral: Tailored behavioral intervention — Participants will receive a standard six session cognitive behavioral intervention for smokeless tobacco cessation combined with supplemental treatment modules based on individual need and preferences.
  Arms: Tailored Intervention
Behavioral: Behavioral activation for elevated depressive symptoms — Participants with elevated depressive symptoms may receive this six session telephone-based behavioral activation intervention.
  Arms: Tailored Intervention
Behavioral: Post-cessation weight gain management — Participants with concerns about gaining weight after quitting smokeless tobacco use may receive this six session telephone-based behavioral self-management intervention designed to help attenuate post-cessation weight gain.
  Arms: Tailored Intervention
Behavioral: Alcohol use risk reduction — Participants engaging in risky alcohol use may receive this six session telephone-based behavioral intervention for reducing alcohol use.
  Arms: Tailored Intervention
Drug: Nicotine replacement therapy - transdermal nicotine patch — Medication selection will be based on individual participant preferences, medical history, and contraindications.
  Other Names: Nicotine patch
  Arms: Tailored Intervention
Drug: Nicotine replacement therapy - nicotine lozenge — Medication selection will be based on individual participant preferences, medical history, and contraindications.
  Other Names: Nicotine lozenge
  Arms: Tailored Intervention
Drug: Nicotine replacement therapy - nicotine gum — Medication selection will be based on individual participant preferences, medical history, and contraindications.
  Other Names: Nicotine gum
  Arms: Tailored Intervention
Drug: Bupropion sustained release — Medication selection will be based on individual participant preferences, medical history, and contraindications.
  Other Names: Zyban
  Arms: Tailored Intervention
Drug: Varenicline — Medication selection will be based on individual participant preferences, medical history, and contraindications.
  Other Names: Chantix
  Arms: Tailored Intervention
Drug: Combination nicotine replacement therapy — Medication selection will be based on individual participant preferences, medical history, and contraindications. Possible combinations include nicotine patch + nicotine lozenge and nicotine patch + nicotine gum.
  Arms: Tailored Intervention
Drug: Combination nicotine replacement therapy + bupropion — Medication selection will be based on individual participant preferences, medical history, and contraindications. Possible combinations include nicotine patch + bupropion, nicotine gum + bupropion, and nicotine lozenge + bupropion.
  Other Names: Medication selection will be based on individual participant preferences, medical history, and contraindications.
  Arms: Tailored Intervention
Behavioral: Tobacco quit line — Referral to the Department of Veterans Affairs tobacco telephone quit line.
  Arms: Facilitated tobacco quit line referral
Behavioral: Educational materials — Information regarding the VA tobacco quit line and associated treatment services, self-help materials for tobacco cessation, and information about tobacco cessation medications available in the VA,
  Arms: Facilitated tobacco quit line referral

SUMMARY:
This is a pilot study designed in an effort to develop and improve access to effective treatments for tobacco use in rural Veterans using a tailored intervention approach. Specifically, we will evaluate a combined behavioral and pharmacological smokeless tobacco cessation which concomitantly addresses comorbid issues commonly experienced by rural tobacco users including elevated depressive symptoms, risky alcohol use, and concerns about weight gain. The objectives are to:

1. Evaluate the feasibility of an individually-tailored telephone intervention for rural smokeless tobacco users
2. Examine the impact of the intervention on treatment utilization, patient satisfaction, and smokeless tobacco cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Use smokeless tobacco on a daily basis
2. Be willing to make a quit attempt in the next 30 days
3. Reside in a rural location
4. Receiving care through the Iowa City VA Health Care System or an affiliated community-based outpatient clinic
5. Able to provide informed consent
6. Telephone access
7. Stable residence

Exclusion Criteria:

1. Planning to move in the next 12 months
2. Terminal illness
3. Unstable psychiatric disorder
4. Incarcerated
5. Institutionalized

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-12; Primary Completion 2019-09 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Treatment satisfaction | Three month follow-up
  Participants' impressions of and satisfaction with their assigned intervention will be assessed via interview.

SECONDARY OUTCOMES:
Tobacco use | Three-and six-month follow-up
  At three- and six-months, participants will be questioned regarding tobacco use over the prior seven days (seven-day point prevalence abstinence). Those reporting abstinence at six-months will be asked to provide a saliva sample for measuring cotinine in order to biochemically verify self-reported tobacco use.
Alcohol use | Three- and six-month follow-up
  Alcohol use during the previous seven days.
Depressive symptoms | Three- and six-month follow-up
  Depressive symptoms will be assessed using the Patient Health Questionnaire 9 (PHQ-9)
Body weight | Three- and six-month follow-up
  Body weight will be assessed via self-report.
Enrollment rate | Six months after study initiation
  The number of participants enrolled will be tracked as a measure of the feasibility of the intervention approach.
Retention | Six months after study initiation
  The proportion of participants who remain in the study throughout the entire six-month study period will be determined as an indicator of the feasibility of the treatment approach.
Treatment attendance | Three-month follow-up
  The number of treatment calls completed at the time of the three-month follow-up assessment will be determined for all participants in the Tailored intervention condition as an indicator of the feasibility of the treatment approach.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Vander Weg, PhD, Principal Investigator — Iowa City VA Health Care System
Locations (1):
- Iowa City VA Healthcare System, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No